CLINICAL TRIAL: NCT04763018
Title: A Randomized Sham Controlled Study of External Neuromodulation to Improve Signs and Symptoms of Dry Eye in Visual Display Terminal Users
Brief Title: Study of External Neuromodulation to Improve Signs and Symptoms of Dry Eye in Visual Display Terminal Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olympic Ophthalmics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLP-OO8
Record Dates: First submitted 2021-02-14; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Visual Display Users With Previously Undiagnosed Dry Eye

STUDY DESIGN:
Intervention Model Description: Day 14-30, all subjects receive therapy device
Who Masked: Participant, Outcomes Assessor
Masking Description: Sham device produces noise but no stimulation energy. Assessor does not know which device the subject received. The subject does not know which device he or she received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Active Comparator): This arm will receive a function iTEAR
  Interventions: Device: iTEAR100
- Sham (Sham Comparator): This arm will receive sham treatment device
  Interventions: Device: iTEAR100

INTERVENTIONS:
Device: iTEAR100 — Neurostimulation external nasal nerve to stimulate tear production

SUMMARY:
Two study arms - sham and treatment; There will be a cross over of the sham group to the treatment group at day 15.

DETAILED DESCRIPTION:
This is a post market study. The active device will be the FDA cleared device used within its labeling. The sham group will receive an iTEAR device which looks identical to and makes noise similar to a fully functional iTEAR device but has a tip that does not vibrate. All subjects in the sham group will crossover to the treatment group after 2 two weeks and all patients will continue to 30 days.

The study will be conducted at up to 5 sites in the United States. It will enroll 30 subjects for 30 days.

This is a double-masked study with 10 subjects receiving sham and 20 subjects receiving treatment. The subjects and the examining investigators are masked to treatment until the crossover.

ELIGIBILITY:
Inclusion Criteria:

* > 6hrs visual display terminal
* OSDI > 13
* One of: SChirmer < 10, One quadrant staining > 2, or Meibomian Gland expression <12

Exclusion Criteria:

* Opinion of investigator that subject not be in the study

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-02-17 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Meibomian Gland change in expressibility | 14 days
  Change in gland expression from meibomian glands
Corneal Staining | 14 days
  Change in Staining of cornea
Basal tear output | 14 days
  Change in the basal output of tears

SECONDARY OUTCOMES:
Safety | 30 days
  Incidence of Events which prevent device usage

CONTACTS AND LOCATIONS:
Locations (1):
- Fishman Vision, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All results will be shared at conclusion of last follow up visit
Supporting Information: Study Protocol, SAP, CSR
Time Frame: December 2021